CLINICAL TRIAL: NCT06230978
Title: Evaluation of a Habit-based Work-up to Support Medication Adherence in Primary Care
Brief Title: Evaluation of a Habit-based Work-up to Support Medication Adherence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Matthew J. Witry, Associate Professor, University of Iowa
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 202311617
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Medication Adherence; Habits
Keywords: Medication adherence; Habit; Medication Beliefs; Pharmacist
MeSH Terms: conditions — Medication Adherence; Habits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): The first 16 patients will receive standard medication counseling from the pharmacist
  Interventions: Behavioral: Standard Medication Counseling
- Habit workup arm (Experimental): The second 16 patients will receive the habit workup in addition to medication counseling
  Interventions: Behavioral: Habit workup; Behavioral: Standard Medication Counseling

INTERVENTIONS:
Behavioral: Habit workup — The patient and pharmacist will work together to specify a cue to help them take their medicine every day (e.g. brushing teeth, getting dressed, eating breakfast, making coffee, alarms, visual reminders etc).
  Arms: Habit workup arm
Behavioral: Standard Medication Counseling — The pharmacist provides standard counseling on the new medication

SUMMARY:
The goal of this clinical trial is to test the impact of a medication-taking habit worksheet and discussion with a pharmacist in patients who are prescribed a new chronic medication for cardiovascular disease or depression. The main questions it aims to answer are:

* What is the feasibility and acceptability of the workup from the perspective of the patients and the clinic?
* What is the impact of the intervention on the formation of medication-taking habits compared to a comparison group who receive standard pharmacist counseling?
* What is the difference in medication adherence beliefs and behaviors for the group receiving the habit workup compared to those receiving standard counseling?

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a habit adherence workup delivered by pharmacy in primary care. The study population will include patients taking new medications for chronic conditions like high blood pressure, high cholesterol, diabetes, and depression.

This study uses a sequential design which involves first evaluating 16 patients without the added habit worksheet, and then the second phase evaluates 16 patients with the habit worksheet. All participants meet with the pharmacist and are provided standard counseling on the new medications. All participants complete the pre and post survey.

The pharmacist will be trained on the medication habit workup worksheet which has the patient choose cues they will use to develop their medication-taking habit. These will include associating the new habit with hygiene habits like toothbrushing, other habits like making coffee or eating breakfast, or visual cues like setting medications out where they will be easily noticed when doing other habits like getting dressed. Patients will take their sheet with them as a reminder of their plan. Patients also will receive medication counseling. The encounters will occur in a private clinic room.

All participants will complete baseline and follow-up surveys, which will include space for open-ended comments.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be fluent to speak and write in English,
* must be prescribed a new chronic medication

Exclusion Criteria:

* Does not manage their own medications independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Report Scale | From enrollment to 100 days following
  Five-items from the medication Adherence Report scale assessed using 5-point Likert scale. Possible range 5-25 (higher values associated with greater medication adherence)
4-item Habit Automaticity Index | From enrollment to 100 days following
  This 4 scale uses four validated items from the Habit Automaticity Index and uses a 5-point Likert scale. Possible range 4-20 (higher values associated with greater automaticity of medication-taking habit)

SECONDARY OUTCOMES:
Beliefs about Medicines Questionnaire | From enrollment to 100 days following
  For this study,, 5 items specific, 5 items general from the beliefs about Medicines questionnaire by Horne. Possible range 5-25 for each scale. (for the specific beliefs, lower values are associated with more positive medication beliefs, with the general, higher numbers are associated with greater medication beliefs)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedar Valley Primary Care & Walk-In Clinic | Waterloo IA, Waterloo, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data on primary and secondary outcomes, and basic demographic information
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year following the close of the study.
Access Criteria: They can email the principle investigator
URL: https://pharmacy.uiowa.edu/people/matthew-witry

REFERENCES:
- [Derived] Witry M, Hoehns J, Phillips LA. Pilot of a pharmacist-delivered habit-based intervention to support medication adherence in primary care. Res Social Adm Pharm. 2026 Jan;22(1):147-151. doi: 10.1016/j.sapharm.2025.09.003. Epub 2025 Sep 6. PMID 40946014